CLINICAL TRIAL: NCT03949517
Title: A Pilot Study of 68Ga PSMA 11 PET/MRI and 68Ga RM2 PET/MRI for Evaluation of Prostate Cancer Response to HIFU Therapy
Brief Title: 68-Ga PSMA 11 PET/MRI and 68-Ga RM2 PET/MRI for Evaluation of Prostate Cancer Response to HIFU Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-48213; PROS0093 (Other: OnCore); IRB-48213 (Other: Stanford IRB)
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BAY 86-7548; gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 68-Ga RM2+68-Ga PSMA11 (Experimental): 68-Ga RM2 first followed by 68-Ga PSMA11 within 2 weeks. Participant will be injected IV with 140 ± 20% mBq of 68-Ga RM2 OR 3 to 7 mCi of 68-Ga PSMA11
  Interventions: Drug: 68-Ga RM2; Drug: 68-Ga PSMA11; Device: Investigational software and coils in PET/MR Scan; Procedure: PET/MRI
- 68-Ga PSMA11+68-Ga RM2 (Experimental): 68-Ga PSMA11 first followed by 68-Ga RM2 within 2 weeks. Participant will be injected IV with 140 ± 20% mBq of 68-Ga RM2 OR 3 to 7 mCi of 68-Ga PSMA11
  Interventions: Drug: 68-Ga RM2; Drug: 68-Ga PSMA11; Device: Investigational software and coils in PET/MR Scan; Procedure: PET/MRI

INTERVENTIONS:
Drug: 68-Ga RM2 — Radioactive agent
  Other Names: 68Ga-DOTA-4-amino-1-carboxymethyl-piperidine-DPhe-Gln-Trp-Ala-Val-Gly-His-Sta-Leu-NH2; 68Ga-DOTA-Bombesin; BAY86-7548
Drug: 68-Ga PSMA11 — Radioactive agent
  Other Names: DFKZ 11; HBED CC PSMA; Heidelberg compound
Device: Investigational software and coils in PET/MR Scan — Investigational software and coils in PET/MR Scan by General Electric Healthcare
Procedure: PET/MRI — Positron emission tomography (PET)/Magnetic resonance imaging (MRI) Scan
  Other Names: Positron emission tomography (PET)/Magnetic resonance imaging (MRI)

SUMMARY:
This study is being conducted to determine whether the combination of imaging agents 68-Ga RM2 and 68-Ga PMSA11 is better at assessing response to high intensity focused ultrasound (HIFU) or high dose rate (HDR) local therapy than standard imaging or biopsy in patients with known prostate cancer.

DETAILED DESCRIPTION:
Primary Objective: To determine feasibility of 68Ga-PSMA-11 PET/MRI and 68Ga-RM2 PET/MRI for evaluation of HIFU or HDR local therapy in patients with known prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Known prostate cancer
* Planned HIFU or HDR local therapy
* Able to provide written consent
* Karnofsky performance status of 50 (or Eastern Cooperative Oncology Group (ECOG) /World Health Organization (WHO) equivalent)

Exclusion Criteria:

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam
* Metallic implants (contraindicated for MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duan H, Ghanouni P, Daniel B, Rosenberg J, Davidzon GA, Aparici CM, Kunder C, Sonn GA, Iagaru A. A Pilot Study of 68Ga-PSMA11 and 68Ga-RM2 PET/MRI for Evaluation of Prostate Cancer Response to High-Intensity Focused Ultrasound Therapy. J Nucl Med. 2023 Apr;64(4):592-597. doi: 10.2967/jnumed.122.264783. Epub 2022 Nov 3. PMID 36328488

RESULTS

PARTICIPANT FLOW:
Groups:
- 68-Ga PSMA11+68-Ga RM2: 68-Ga PSMA11 first followed by 68-Ga RM2 within 2 weeks, then receive high-intensity focused ultrasound (HIFU). Participant will be injected IV with 140 ± 20% mBq of 68-Ga RM2 OR 3 to 7 mCi of 68-Ga PSMA11
- 68-Ga RM2+68-Ga PSMA11: 68-Ga RM2 first followed by 68-Ga PSMA11 within 2 weeks, then receive HIFU. Participant will be injected IV with 140 ± 20% mBq of 68-Ga RM2 OR 3 to 7 mCi of 68-Ga PSMA11
Period: Pre-HIFU Period, Imaging Timepoint 1
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Pre-HIFU Period, Imaging Timepoint 2
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: HIFU Treatment
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Post-HIFU Period, Imaging Timepoint 1
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Post-HIFU Period, Imaging Timepoint 2
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 68-Ga PSMA11+68-Ga RM2 | 68-Ga RM2+68-Ga PSMA11 | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.5) | 63.9 (8.1) | 64.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which an Assessment of PET Based Therapeutic Response to HIFU is Successfully Obtained
Description: Positron emission tomography (PET) based of Assessment of Local Therapeutic Response. Therapeutic response to HIFU will be assessed by 68-Ga PSMA 11 and 68-Ga RM2 PET scans.
Time Frame: Up to approximately 2 hours to complete each scan
Measure: Count of Participants; unit: Participants
Groups:
- 68-Ga PSMA11: 68-Ga PSMA11 scan before and after HIFU
- 68-Ga RM2: 68-Ga RM2 scan before and after HIFU
Arm/Group | 68-Ga PSMA11 | 68-Ga RM2
Number analyzed (Participants) | 14 | 14
Participants | 14 | 14

ADVERSE EVENTS:
Time Frame: 4 weeks, plus safety follow up at up to 72 hours after the final scan
Arm/Group | 68-Ga PSMA11 | 68-Ga RM2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03949517/Prot_SAP_002.pdf